CLINICAL TRIAL: NCT04367701
Title: Congenital Heart Surgery in Pediatric Patients With Beta-Thalassemia Major : Analysis of Hemolysis During Cardiopulmonary Bypass
Brief Title: Congenital Heart Surgery in Pediatric Patients With Beta-Thalassemia Major
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, simon Halim Armanious, Lecturer, Ain Shams University
Other Study IDs: Thalassemia CHD
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Hemolysis
MeSH Terms: conditions — Hemolysis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Thalassemia group: 16 pediatric patients with thalassemia major undergoing surgery for repair of congenital heart disease.
  Authors measure hemolysis by free plasma hemoglobin concentration.
  Interventions: Diagnostic Test: Hemolysis
- Control group: 25 pediatric patients with demographic data related to those in thalassemia group, undergoing surgery for repair of congenital heart disease.
  Authors measure hemolysis by free plasma hemoglobin concentration
  Interventions: Diagnostic Test: Hemolysis

INTERVENTIONS:
Diagnostic Test: Hemolysis — Authors measured free plasma hemoglobin concentration in gram

SUMMARY:
Authors compared incidence of Hemolysis on Cardiopulmonary Bypass surgery for repair of congenital heart disease in Pediatric Patients between patients with thalassemia major and control group

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Patients with thalassemia major.
* Pediatric Patients with congenital heart disease undergoing surgical repair.

Exclusion Criteria:

* known hepatic or renal disease
* uncontrolled active hemolytic reaction
* emergency surgery
* redo surgery

Ages: 6 Months to 12 Years | Sex: All
Age Groups: Child
Study Population: Patients with thalassemia major undergoing surgical repair for congenital heart disease
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2012-01-15 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Hemolysis | 3 hours
  Authors measure hemolysis by free plasma hemoglobin concentration

CONTACTS AND LOCATIONS:
Overall Officials: Galal Mo El kadi, Doctor, Study Chair — Professor

IPD SHARING:
Plan to Share IPD: No